CLINICAL TRIAL: NCT06864065
Title: Study of Emotional Regulation and Underlying Prefrontal Activity in Binge Eating Disorder
Acronym: EmoBED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: INSERM UMR 1322 LINC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/886
Record Dates: First submitted 2025-02-11; First posted 2025-03-07 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Binge-Eating Disorder; Emotional Eating; Healthy Volunteers
Keywords: Binge-Eating Disorder; Emotion regulation; fNIRS; Prefrontal cortex; Eating disorder; Emotional Eating
MeSH Terms: conditions — Binge-Eating Disorder; Emotional Eating; Emotional Regulation; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: It is important to note that no drugs are tested. The task (emotion regulation) is consistent for all groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with binge eating desorders (Experimental): Patients with binge eating desorders
  Interventions: Behavioral: Emotion regulation task (fNIRS recording during the emotional regulation task)
- healthy volunteers with a low score at the emotion eating scale compare to median (Experimental): group matched with patients for age and body mass index
  Interventions: Behavioral: Emotion regulation task (fNIRS recording during the emotional regulation task)
- healthy volunteers with a high score at the emotion eating scale compare to median (Experimental): group matched with patients for age and body mass index
  Interventions: Behavioral: Emotion regulation task (fNIRS recording during the emotional regulation task)
- healthy volunteers normo-weight group with a low score at the emotion eating scale compare to median (Experimental): healthy volunteers with normo-weight group matched with patients only in age but not in Body Mass Iindex with an Emotional Eating score below the median
  Interventions: Behavioral: Emotion regulation task (fNIRS recording during the emotional regulation task)

INTERVENTIONS:
Behavioral: Emotion regulation task (fNIRS recording during the emotional regulation task) — No drugs were used in this study. All participants perform an emotion regulation task. More precisely, they have to down regulate negative emotions elicited by negative pictures using a cognitive reaprasal strategy. To this end, they have to change the meaning of the picture they are watching in order to decrease motional intensity.

SUMMARY:
The goal of this exploratory, interventional, multicentre study is to compare the prefrontal activity during a negative emotion regulation task in women with Binge-Eating Disorder (BED) and healthy women with and without Emotional Eating (EE).

The aim of this study is to compare the prefrontal processing of cognitive control of emotions between BED and EE and to compare the emotional processing and emotional experience between BED and EE.

The study will thus compare four experimental groups: patients with BED, BMI-matched healthy volunteers with EE, BMI-matched healthy volunteers, and healthy volunteers of normal weight without BED.

Participants will perform a down-regulation task of negative emotions elicited by negative pictures. During this task, their cerebral activity will be recorded using functional near-infrared spectroscopy (fNIRS), as well as their autonomous activity (skin conductance, pulse rate, respiration rate).

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 60 years old (including 60)
* Right-handed.
* For patients only : diagnosed with Binge Eating Desordors according to DSM criteria.
* Membership of a French social security scheme or beneficiary of such a scheme.
* Non-opposition of the subject to participate in the study.

Non inclusion Criteria:

Healthy volunteers only :

* Suffering from an eating disorder or any other psychiatric disorder.
* History of bariatric surgery.

All subjects (healthy volunteers and patients) :

* Rare obesity (genetic or syndromic).
* Specific addictions (substances or behaviors).
* Neurological disorders and/or history of stroke or head trauma.
* Presence of lesions, wounds or dermatitis at the sites where the recording devices are applied.
* Any serious acute or chronic illness other than the pathology under study, or any treatment likely to interfere with the evaluation of the parameter under study.
* Inability to follow protocol requirements.
* Subject unlikely to cooperate with the study and/or poor cooperation anticipated by the investigator.
* Subject unable to speak French and/or unable to read.
* Pregnant or breast-feeding women.
* Persons deprived of their liberty by judicial or administrative decision; persons under compulsory psychiatric care; persons admitted to a health or social institution for purposes other than research.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of prefrontal cortex activity using functional near-infrared imaging (fNIRS). | Day 1 during the viewing of images with negative valence
  The fNIRS signal represents the concentration of oxyhemoglobin and deoxyhemoglobin over time. It provides information about the local oxygen demand of the brain and therefore its activity.
  It is these concentrations during the regulatory task that are used as the primary outcome measure.

SECONDARY OUTCOMES:
Psychophysiological measurements: electrodermal activity | Day 1 during the viewing of images with negative valence
  Skin conductance measures are recorded These provide information on the autonomic nervous system (sympathetic and parasympathetic) and thus on emotional processing and arousal.
Psychophysiological measurements: electrocardiogram | Day 1 during the viewing of images with negative valence
  Electrocardiogram measures are recorded These provide information on the autonomic nervous system (sympathetic and parasympathetic) and thus on emotional processing and arousal.
Psychophysiological measurements: respiratory rate | Day 1 during the viewing of images with negative valence
  Respiratory rate is recorded These provide information on the autonomic nervous system (sympathetic and parasympathetic) and thus on emotional processing and arousal.

CONTACTS AND LOCATIONS:
Overall Officials: AMSALLEM Anne-Cécile, MD, Study Director — CHU de Besançon
Locations (3):
- France (3):
  - UFC - UFR Santé, Besançon
  - CHU de Besançon, Besançon
  - CHU de Dijon, Dijon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parker MN, Burton Murray H, Piers AD, Muratore A, Lowe MR, Manasse SM, Ayaz H, Juarascio AS. Prefrontal cortex activation by binge-eating status in individuals with obesity while attempting to reappraise responses to food using functional near infrared spectroscopy. Eat Weight Disord. 2023 Mar 30;28(1):34. doi: 10.1007/s40519-023-01558-z. PMID 36995567
- [Background] Dingemans A, Danner U, Parks M. Emotion Regulation in Binge Eating Disorder: A Review. Nutrients. 2017 Nov 22;9(11):1274. doi: 10.3390/nu9111274. PMID 29165348
- [Background] Arexis M, Feron G, Brindisi MC, Billot PE, Chambaron S. A scoping review of emotion regulation and inhibition in emotional eating and binge-eating disorder: what about a continuum? J Eat Disord. 2023 Nov 10;11(1):197. doi: 10.1186/s40337-023-00916-7. PMID 37950264